CLINICAL TRIAL: NCT04741373
Title: Study on Pulmonary Rehabilitation Intervention Including Oral Nutritional Supplements(ONS) on Stable COPD Patients Who Are Under Nutrition
Brief Title: Study on Pulmonary Rehabilitation for Stable Chronic Obstructive Pulmonary Disease(COPD) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Huadong Hospital to Fudan
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Nutritional Support; Aerobic Exercise; Respiratory Function Tests; Body Composition; Muscle Strength
Keywords: oral nutritional supplements; aerobic exercise; resistance exercise; respiratory function tests; body composition
MeSH Terms: interventions — Dietary Supplements; Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group of health education (Placebo Comparator)
  Interventions: Other: health education
- Group of health education and rehabilitation exercise (Active Comparator)
  Interventions: Behavioral: rehabilitation exercise; Other: health education
- Group of health education,exercise and ONS (Experimental)
  Interventions: Dietary Supplement: oral nutritional supplements; Behavioral: rehabilitation exercise; Other: health education

INTERVENTIONS:
Dietary Supplement: oral nutritional supplements — oral nutritional supplements, 400-600kcal/day;
  Arms: Group of health education,exercise and ONS
Behavioral: rehabilitation exercise — Aerobic exercise: fixed cycling in rehabilitation center or walking at home, 3-5 times/week, Resistance exercise: lift dumbbell by upper limb, raise legs tying sandbags, 2-3 times/week
  Arms: Group of health education and rehabilitation exercise; Group of health education,exercise and ONS
Other: health education — Establish WeChat group or QQ group or telephone contact, and regularly distribute electronic science pictures or small videos

SUMMARY:
To compare the difference of effectiveness for stable COPD patients with poor nutritional status among three groups named health education, upper and lower limb exercises, and oral nutritional supplements. Then formulate the best pulmonary rehabilitation guidance strategy according to the result of this trial.

DETAILED DESCRIPTION:
This study is a clinical randomized, non-blinded, controlled study in China. The participants will be 90 stable COPD patients with poor nutritional status selected by the community or primary hospitals. On the principle of having no statistical difference in indicators such as baseline age, Global Initiative for Chronic Obstructive Lung Disease（GOLD） staging, and medication oxygen consumption among the groups , the trial will randomly be divided into three groups: health education group, health education + upper and lower extremity exercise group, health education + upper and lower extremity exercise + oral nutritional supplements group.

A 12-week pulmonary rehabilitation clinical study will be conducted to observe the difference of outcome indicators among the three groups like nutritional status (24hr diet, body weight, body composition, albumin), pulmonary function (classification and staging), muscle strength and muscular endurance (grip strength, 6-minute walking distance(6MWD)), inflammation factors and St. George's Respiratory Questionnaire (SGRQ) score. Moreover outcome indicators after 24 weeks like patient weight, SGRQ score and GOLD staging also will be recorded for comparison.

The project will evidence-based provide effective means like nutrition and exercise for Chinese malnourished COPD patients who are at stable stage. And popular science books on pulmonary rehabilitation based on this trial will be compiled to record the best pulmonary rehabilitation guidance strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate and severe COPD with a clear diagnosis of lung function, (moderate-forced expiratory volume at one second（FEV1）/forced vital capacity（FVC）<0.7, FEV1% between 50-80%; severe-FEV1/FVC<0.7, FEV1% < 50%).
2. Patients are at stable stage of COPD which means hospital admission <2 times due to acute exacerbation in the past two years, no changes in respiratory symptoms and medication in the past month.
3. Patients have not participated in any form of pulmonary rehabilitation in the past at least 0.5 year and simultaneously have not taken any form of nutritional supplements in the past at least 2 weeks.
4. Malnutrition criteria: Mini Nutritional Assessment-ShortForm(MNA-SF) ≤ 12 points; or Body Mass Index(BMI) ≤ 21kg/m2.
5. Volunteers have the ability to complete the test of lung function, grip strength, 6MWD, body composition and blood index tests.

Exclusion Criteria:

1. Patients suffer from significant diseases which will cause the subjects to be at risk due to participating in the research, or affect the research results and the subjects' ability to participate in the research,including severe diseases of liver and kidney, nervous system, endocrine and digestive system .
2. Patients have ischemic heart disease with a history of angina pectoris, or uncontrolled chest tightness and angina pectoris after activities recently.
3. Patients have severe pulmonary hypertension or grade IV by heart function grade of New York Heart Association(NYHA).
4. Arterial oxygen saturation (SpO2) <88% or PaCO2> 55mmHg in a quiet state.
5. Those whose life cycle is expected to be less than 6 months.
6. Walking restriction is limited in 300m because of intermittent claudication caused by peripheral arterial disease or osteoporosis.
7. Patients lost capability of autonomous activity or have cognitive impairment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Weight | three months
  Anthropometry
Fat free mass | three months
  Anthropometry
Fat mass | three months
  Anthropometry
Muscle mass | three months
  Anthropometry

SECONDARY OUTCOMES:
Grip strength | three months
  Muscle strength
6MWD | three months
  Muscle endurance strength

CONTACTS AND LOCATIONS:
Overall Officials: Jie Chen, PhD, Study Director — Huadong Hospital
Locations (1):
- Huadong Hospital Affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No